CLINICAL TRIAL: NCT04213391
Title: Randomized,Double-blind, Placebo-controlled, Efficacy and Safety Study of Sulforaphane in Patients With Prodromal to Mild Alzheimer's Disease
Brief Title: Effects of Sulforaphane in Patients With Prodromal to Mild Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Wulab-AD sulforaphane
Record Dates: First submitted 2019-11-13; First posted 2019-12-30 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sulforaphane group (Experimental): The patients will take sulforaphane for 24 weeks, 2550mg once a day.
  Interventions: Dietary Supplement: sulforaphane
- Placebo group (Placebo Comparator): The patients will take placebo for 24 weeks, 2550mg once a day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: sulforaphane — Sulforaphane take 2550mg once a day.
  Arms: sulforaphane group
Dietary Supplement: Placebo — Placebo take 2550mg once a day.
  Arms: Placebo group

SUMMARY:
In this proposed study, the investigators will evaluate the efficacy, safety and related mechanism of sulforaphane in treatment of Alzheimer's disease (AD). The study will recruit 160 AD patients, and then these patients will be randomized to sulforaphane group or placebo group (80 patients per arm) for 24 weeks clinic trial. Clinical efficacy and safety assessment will be done at screen/baseline, 4 week, 12 week, and 24 week. The specific aims are to compare sulforaphane versus placebo on: clinical core symptoms; biological samples also will be collected, and stored to research related mechanisms. During the study period, safety index including blood and urine routine, liver and kidney function, coagulation index and clinical effect index about neuropsychological scales will be recorded.

DETAILED DESCRIPTION:
In this proposed study, the investigators will evaluate the efficacy, safety and related mechanism of sulforaphane in treatment of AD. The study will recruit 160 AD patients, then these patients will be randomized to sulforaphane group or placebo group (80 patients per arm) for 24 weeks clinic trial. Clinical efficacy and safety assessment will be done at screen/baseline, 4 week, 12 week, 24 week. The specific aims are to compare sulforaphane versus placebo on: 1) clinical core symptoms; The investigators hypothesize that (1) sulforaphane is superior to placebo in the treatment of clinical symptoms in patients with AD, measured by the ADAS-cog, MMSE Scale, Moca; (2) Biological samples will be collected, and stored so that the hypothesis sulforaphane may alter oxidative stress indexes or inflammatory biomarkers, and influence histone deacetylase inhibitor mechanism or inflammatory mechanism et al that may be significantly correlated with clinical improvement. (3) Safety index including blood and urine routine, liver and kidney function, coagulation index and clinical effect index about neuropsychological scales will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range from 50 to 75 (including 50 and 75 years old), regardless of ethnic group or gender;
* 2. The subjects should be able to complete the cognitive ability measurement and other tests specified in the protocol;
* 3. Meeting the criteria for likely Alzheimer's Disease （AD） dementia (2011) by National Institute of Neurological Disorders and Strokes - Alzheimer's Disease and Related Diseases Association（NINCDS-ADRDA）;
* 4. Patients with mild dementia: the total score of Mini-Mental State Examination (MMSE) : ≥22 points; Clinical Dementia Rating scale （CDR）score > or equal to 0.5 and < or equal to1；The MMSE score provides evidence of mild disease severity and the CDR-GS score indicates that the patients have noticeable amnestic (pAD) or cognitive and functional (mAD) deficits
* 5. The total score of the Hachinski Ischemic Score （HIS ）was < 4.
* 6. Hamilton depression scale (17 items) total score ≤7 points;
* 7. Brain MRI shows a high likelihood of AD;
* 8. Before enrollment, patients should take a stable dose of dementia drugs (donepezil 5mg) ≥8 weeks;
* 9. The expected survival time is > 1 year;
* 10. Subjects should have a stable and reliable caregiver, or at least have frequent contact with the caregiver (at least 3 days per week and at least 2 hours per day), who will help patients participate in the whole study; Caregivers must accompany the subjects to the visit and assist in completing the relevant scale.

Exclusion Criteria:

* 1. Refuse to sign the inform consent form;
* 2. Other causes of dementia: known vascular, central nervous system infection ,Parkinson's disease, traumatic brain dementia, other physical and chemical factors; serious body disease , intracranial space-occupying lesions, endocrine system disease, such as thyroid disease, and a lack of vitamin B12, folic acid, or any other known causes of dementia.
* 3. Central nervous system diseases (including stroke, optic neuromyelitis, Parkinson's disease, epilepsy, etc.);
* 4. Obvious positive signs of nervous system examination;
* 5. Psychotic patients, including schizophrenia or other disorders with bipolar disorder, major depression or delirium;
* 6. Uncontrolled hypertension or hypotension during screening: systolic blood pressure ≥180（millimetres of mercury ）mmHg or < 90mmhg, or diastolic blood pressure ≥120mmHg or < 60mmhg;
* 7. Unstable or severe diseases of the heart, lung, liver, kidney and hematopoietic system according to the judgment of the researchers;
* 8. Patients with incurable visual and auditory disorders that cannot complete neuropsychological tests and scales;
* 9. Female subjects who are positive in pregnancy test or breast-feeding and who cannot take effective contraceptive measures or have a birth plan;
* 10. Severe allergy, non-allergic drug reaction or multi-drug allergy history;
* 11. Participated in other clinical trials within 3 months before screening visit;
* 12. Taking any health care products related to brain and brain improvement currently and failing to keep the promise to stop using the above products;
* 13. Other conditions are unsuitable for participating in this study according to the judgement of researchers.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-05-10 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The Alzheimer's Disease Assessment Scale | From baseline to 24 weeks
  The Alzheimer's Disease Assessment Scale (ADAS-cog) will be performed to test the cognition of patients at the enrollment, week 12 and week 24. The score ranges from 0 to 75，and higher values represent a better outcome.

SECONDARY OUTCOMES:
Alzheimer's Disease Collaborative research group-Activities of Daily Living scores. | From baseline to 24 weeks
  Alzheimer's Disease Collaborative research group-Activities of Daily Living scores (ADCS-ADL) will be performed to test the activities of patients at the enrollment,week 6 and week12.The score ranges from 0 to 54，and higher values represent a better outcome.
Neuropsychiatric Inventory scores | baseline time to 24 weeks
  Neuropsychiatric Inventory scores (NPI) will be performed to test the mental symptoms of patients at the enrollment and week12.The score ranges from 0 to 144，and higher values represent a worse outcome.
Mini-Mental State Examination scores | baseline time to 24 weeks
  Mini-Mental State Examination scores(MMSE) will be performed to test the cognition of patients at the enrollment and week12.The score ranges from 0 to 30，and higher values represent a better outcome.
Montreal Cognitive Assessment scores | baseline time to 24 weeks
  Montreal Cognitive Assessment scores (MoCA) will be performed to test the cognition of patients at the enrollment and week12.The score ranges from 0 to 30，and higher values represent a better outcome.
Clinician Interview-Based Impression of Change plus caregiver input | baseline time to 24 weeks
  Clinician Interview-Based Impression of Change plus caregiver input (CIBIC-plus) is widely used in antidementia drug trials. It comprises Likert scales for disease severity and changes, and written accounts summarizing semistructured interviews evaluating behavior, cognition, and function.

OTHER OUTCOMES:
Oxidative stress indexes | At baseline and 24 week/endpoint
  The change of Oxidative stress indexes as tested by Oxidative stress indexes detection kit
Epigenetics indicators | At baseline and 24 week/endpoint
  The change of Epigenetics indicators as tested by Epigenetics indicators
Cytokines & Chemokines | At baseline and 24 week/endpoint
  The change of Cytokines & Chemokines as tested by Cytokines & Chemokines detection kit
Metabolites | At baseline and 24 week/endpoint
  The change of Metabolites as tested by Metabolites detection kit
RNA expression | At baseline and 24 week/endpoint
  The change of RNA expression as tested by RNA expression detection kit
Intestinal microflora | At baseline and 24 week/endpoint
  The change of intestinal microflora as tested by Metagenomic technique

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee S, Choi BR, Kim J, LaFerla FM, Park JHY, Han JS, Lee KW, Kim J. Sulforaphane Upregulates the Heat Shock Protein Co-Chaperone CHIP and Clears Amyloid-beta and Tau in a Mouse Model of Alzheimer's Disease. Mol Nutr Food Res. 2018 Jun;62(12):e1800240. doi: 10.1002/mnfr.201800240. Epub 2018 May 28. PMID 29714053
- [Background] Hou TT, Yang HY, Wang W, Wu QQ, Tian YR, Jia JP. Sulforaphane Inhibits the Generation of Amyloid-beta Oligomer and Promotes Spatial Learning and Memory in Alzheimer's Disease (PS1V97L) Transgenic Mice. J Alzheimers Dis. 2018;62(4):1803-1813. doi: 10.3233/JAD-171110. PMID 29614663
- [Background] Jhang KA, Park JS, Kim HS, Chong YH. Sulforaphane rescues amyloid-beta peptide-mediated decrease in MerTK expression through its anti-inflammatory effect in human THP-1 macrophages. J Neuroinflammation. 2018 Mar 12;15(1):75. doi: 10.1186/s12974-018-1112-x. PMID 29530050
- [Background] Kim J, Lee S, Choi BR, Yang H, Hwang Y, Park JH, LaFerla FM, Han JS, Lee KW, Kim J. Sulforaphane epigenetically enhances neuronal BDNF expression and TrkB signaling pathways. Mol Nutr Food Res. 2017 Feb;61(2). doi: 10.1002/mnfr.201600194. Epub 2016 Nov 30. PMID 27735126
- [Background] Zhao F, Zhang J, Chang N. Epigenetic modification of Nrf2 by sulforaphane increases the antioxidative and anti-inflammatory capacity in a cellular model of Alzheimer's disease. Eur J Pharmacol. 2018 Apr 5;824:1-10. doi: 10.1016/j.ejphar.2018.01.046. Epub 2018 Jan 31. PMID 29382536
- [Background] Zhang R, Zhang J, Fang L, Li X, Zhao Y, Shi W, An L. Neuroprotective effects of sulforaphane on cholinergic neurons in mice with Alzheimer's disease-like lesions. Int J Mol Sci. 2014 Aug 18;15(8):14396-410. doi: 10.3390/ijms150814396. PMID 25196440